CLINICAL TRIAL: NCT01450878
Title: Interest of a High Dose of Erythropoietin Administered During Graft Processing for Early Graft Outcome in Kidney Transplant Recipients.
Brief Title: Renal Graft Function After Treatment With Erythropoietin (EPO)
Acronym: FRETEP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of patients eligible for the study.
Sponsor: University Hospital, Limoges (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I09002 FRETEP
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Ischemia
Keywords: high dose of EPO; transplant kidney; cadaveric organ donor; mono-organ (kidney) retrieval; patient; kidney graft
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Graft with EPO (Experimental): intravenous 1000 000UI beta-epoietin one hour before organe retrieval.
  Interventions: Drug: beta-epoietin
- graft without EPO (No Intervention): no injection befoe organ retrieval

INTERVENTIONS:
Drug: beta-epoietin — 100 000UI beta-epoietin injection one hour before organ retrieval
  Arms: Graft with EPO

SUMMARY:
Background : Numerous studies have outlined the cellular pleiotropic effects of erythropoietin (EPO) and their role in the prevention of ischemic-reperfusion lesion such as after acute ischemic injury of the brain or the heart. However, most of these studies were carried out in animal models and no definitive proof exists today to demonstrate that EPO has similar beneficial effects in human pathology.

Purpose : The aim of the study is to demonstrate that in humans, EPO can protect against ischemic-reperfusion lesions in a model of ischemia i.e. kidney transplantation.

DETAILED DESCRIPTION:
Abstract : Since the discovery that EPO and its receptor are expressed in various tissues, numerous studies have demonstrated that EPO is not only involved in erythropoiesis but also exerts pleiotropic effects on cells. Among these, one of the most exciting is its role in the prevention of ischemic-reperfusion lesions such as after acute ischemic injury of the brain or the heart. However, most of these studies were carried out in animal models and no definitive proof exists today to demonstrate that EPO has similar beneficial effects in human pathology. Kidney transplantation is one ischemic situation where EPO pleiotropic effects could be of great interest since ischemic-reperfusion lesions have been involved in delayed graft function and impaired graft outcomes.

The aim of this prospective randomized double blind study is to assess the effect of 100 000 UI of béta-epoiétin on kidney graft function, given to the deceased donor one hour before the retreaval of the organ. Recipients will be followed for three months in order to evaluate kidney function (glomerular filtration rate) and the number of acute rejection episodes to determine whether beta-epoietin could modify the immunogenicity of the graft.

ELIGIBILITY:
Inclusion Criteria:

* donor:

  * cadaveric organ donor,
  * age ≥ 18 years,
  * mono-organ (kidney) retrieval,
  * retrieval done in the centres of Limoges, Bordeaux, Toulouse, Angers, Brest, Nantes, Poitiers, Rennes, Tours,
  * hematocrit ≤ 45%.
* Recipient:

  * age ≥ 18 years,
  * on the waiting list for a kidney graft.

Exclusion Criteria:

* living donors,
* age under 18 years,
* multi-organ retrieval,
* donor hematocrit above 45%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
a plasma creatinin level | 5 days
  To assess the effect of an injection of 100 000 UI of beta-epoitein during graft processing, on the proportion of renal recipients with a plasma creatinin level below 250 µM at day 5 after transplantation in the absence of hemodialysis, death or transplantectomy.

SECONDARY OUTCOMES:
The incidence of delayed graft function defined as follows: | 48 hours
  The incidence of delayed graft function defined as follows: combination of the need for dialysis (except dialysis for hyperkalemia or volume overload) or creatinine reduction ratio of less than 25% within the first 48 h post-transplant.
MDRD glomerular filtration rate at one and three months | three months
  MDRD glomerular filtration rate at one and three months
The incidence of acute rejection during the first three months | three months
  The incidence of acute rejection during the first three months

CONTACTS AND LOCATIONS:
Overall Officials: Marie ESSIG, MD, Principal Investigator — CHU LIMOGES
Locations (18):
- France (18):
  - Néphrologie, Angers
  - CHU d'ANGERS - CHPOT, Angers
  - CHU de BORDEAUX - CHPOT, Bordeaux
  - CHU de BORDEAUX - Service de Néphrologie, Bordeaux
  - Néphrologie, Brest
  - CHU de BREST - CHPOT, Brest
  - CHU de LIMOGES - CHPOT, Limoges
  - CHU de LIMOGES - Service de Néphrologie, Limoges
  - CHU de NANTES - CHPOT, Nantes
  - CHU de NANTES - Service de Néphrologie, Nantes
  - Néphrologie, Poitiers
  - CHU de POITIERS - CHPOT, Poitiers
  - CHU de RENNES - CHPOT, Rennes
  - CHU de RENNES - Service de Néphrologie, Rennes
  - CHU de TOULOUSE - CHPOT, Toulouse
  - CHU de TOULOUSE - Service de Néphrologie, Toulouse
  - Néphrologie, Tours
  - CHU de TOURS - CHPOT, Tours